CLINICAL TRIAL: NCT06185998
Title: Impact of the Nature and Interface of the Tracheostomy Cannula on Dyspnea in Patients Weaning From Artificial Ventilation in Weaning Unit
Acronym: DYSTRACH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: APHP230863
Record Dates: First submitted 2023-11-23; First posted 2023-12-29 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2023-12

CONDITIONS: Prolonged Weaning
Keywords: prolonged weaning; tracheostomy; dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plated balloon tracheostomy cannulas (Experimental): 4 interfaces are tested: cap, ventilator, filter and phonation valve
  Interventions: Device: low pressure tracheostomy cannulas; Device: plated balloon tracheostomy cannulas
- low pressure balloon tracheotomy cannulas (Active Comparator): 4 interfaces are tested: cap, ventilator, filter and phonation valve
  Interventions: Device: low pressure tracheostomy cannulas; Device: plated balloon tracheostomy cannulas

INTERVENTIONS:
Device: low pressure tracheostomy cannulas — The tracheostomy tube is changed according to the randomization sequence, a filter is connected for 5 minutes; then baseline data will be assessed. The tracheostomy tube is then connected to the four interfaces for 30 minutes each. Parameters is measured after each 30-minute period. The cuff of the tracheostomy tube will be deflated using a syringe when the interface is a filter, phonation valve, or cap. In contrast, the cuff will be inflated when the interface is the ventilator.
  The cuff is inflated with a manometer for the low-pressure balloon tracheostomy tube and with the minimum and sufficient amount of injectable water for the plated balloon tracheostomy tube to avoid overpressure
  Other Names: non fenestrated TRACOE® twist; TRACOE tracheostomy tubes with low-pressure cuff; low wall thickness and a good fit of the inner cannula in the outer cannula
Device: plated balloon tracheostomy cannulas — The tracheostomy tube is changed according to the randomization sequence, a filter is connected for 5 minutes; then baseline data will be assessed. The tracheostomy tube is then connected to the four interfaces for 30 minutes each. Parameters is measured after each 30-minute period. The cuff of the tracheostomy tube will be deflated using a syringe when the interface is a filter, phonation valve, or cap. In contrast, the cuff will be inflated when the interface is the ventilator.
  The cuff is inflated with a manometer for the low-pressure balloon tracheostomy tube and with the minimum and sufficient amount of injectable water for the plated balloon tracheostomy tube to avoid overpressure
  Other Names: Bivona® TTS™ Tracheostomy Tubes; silicone tube TTS™ cuff; tubes are coated with a SuperSlick®; soft, confort and flexible tube

SUMMARY:
This trial aims to assess dyspnea intensity in tracheostomized patients undergoing prolonged artificial ventilation weaning. The primary outcome is dyspnea measured by the Visual Analogue Scale (VAS-Dyspnea). A comparison between low-pressure balloon tracheostomy cannula and plated balloon cannula and four interfaces (Cap, ventilator, phonation valve, or filter) are tested. The secondary outcomes including Multidimensional Dyspnea Profile, pain, anxiety VAS, and tolerance under different interfaces. The multicenter, cross-over study involves 76 patients over 25 months, each serving as their own control. Cap is always evaluated first but the order of the three interfaces (ventilator, phonation valve, or filter) and type of cannula are chosen by randomization. The study is conducted in three weaning centers (SRPR units) at Pitié-Salpêtrière, Bligny, and Forcilles.

DETAILED DESCRIPTION:
Dyspnea is common in patients ventilated in intensive care and SRPR units, and it can generate states of post-traumatic stress. Due to the prolonged duration of artificial ventilation, tracheostomized patients, for the purpose of prolonged weaning from artificial ventilation, are particularly exposed to dyspnea.

The main objective is to compare the respective impact of a low-pressure balloon tracheostomy cannula and a plated balloon cannula on the dyspnea intensity of tracheostomized patients in spontaneous ventilation, with the cannula closed by a cap. The primary outcome is the Visual Analogue Scale (VAS) for dyspnea (VAS-Dyspnea).

The investigators will compare low pressure versus plated balloon tracheostomy cannulas, considering the sensory and emotional components of dyspnea, as well as tolerance, pain, comfort, and anxiety under four different interfaces: ventilator, phonation valve, Cap, or filter. This will be measured through the following secondary outcomes:

* VAS-Dyspnea
* Multidimensional Dyspnea Profile
* Pain and anxiety VAS This multicenter study (SRPR Pitié-Salpêtrière, Bligny, and Forcilles) will be randomized in a cross-over design, comparing the use of two types of low-pressure or plated balloon cannulas over two consecutive days. For each cannula, four interfaces will be connected in a row starting with the cap. The order in which the other three interfaces will be set up will be randomized (ventilator, filter, and phonation valve).

It is a cross-over including 76 patients, with each serving as their his own control, over 25 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient admitted to SRPR with respiratory and hemodynamic stability
* Patient with a tracheostomy tube
* Deflated balloon for more than 6 hours per day
* Able to tolerate at least 1 hour on cap and phonation valve (deflated balloon)
* Able to remain at least 3 consecutive hours without ventilation
* Patient with at least one non-zero dyspnea numerical rating scale (NRS) score in the 72 hours preceding inclusion
* Able to respond to self-administered questionnaires on dyspnea
* Patients affiliated with a social security system or beneficiaries of such a system (excluding State Medical Assistance)
* Patients who have given their informed consent
* No significant expected changes in the administration of anxiolytic and analgesic treatments with anti-dyspneic properties within 2 days

Exclusion Criteria:

* Pregnant women (verified by a blood or urine test during hospitalization for all women of childbearing age)
* Patients deprived of liberty or under legal protection (guardianship or curatorship)
* Patients unable to consent to the research
* Contraindication to the use of a 7 mm tracheostomy tube
* Patient presenting the combination of major swallowing disorders and excessive salivary secretion making the deflation of the tracheostomy tube balloon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Dyspnea visual analogic scale (VAS) with cap | 30 minutes after using each interfaces
  The VAS of dyspnoea evaluate the severity of dyspnoea, the index has 10 numerical values, rated on a scale from 0-10, each value corresponding to an intensity of breathlessness. It is an easy-to-use scale for patients.

SECONDARY OUTCOMES:
Dyspnea visual analogic scale (VAS) after 30 min breathing with filter, ventilator and phonation valve | 30 minutes after using each interfaces
  The VAS of dyspnoea evaluate the severity of dyspnoea, the index has 10 numerical values, rated on a scale from 0-10, each value corresponding to an intensity of breathlessness. It is an easy-to-use scale for patients.
Multidimensional Dyspnea Profile (MDP) | 30 minutes after using each interfaces
  The Multidimensional Dyspnea Profile (MDP) assesses overall breathing discomfort, sensory qualities, and emotional responses
Biological variable : Heart rate | 30 minutes after using each interfaces
  Heart rate (beat per minute)
Biological variable : Respiratory rate | 30 minutes after using each interfaces
  Respiratory rate (cycles per minute)
Biological variable : Systolic and diastolic systemic blood pressure | 30 minutes after using each interfaces
  Systolic and diastolic systemic blood pressure (millimeters of mercury - mmHg)
Biological variable : Pulsed oxygen saturation | 30 minutes after using each interfaces
  Pulsed oxygen saturation (percentage %)
Pain visual analogic scales (VAS) | 30 minutes after using each interfaces
  evaluate the severity of pain the index has 10 numerical values, rated on a scale from 0-10, each value corresponding to an intensity pain and anxiety. It is an easy-to-use scale for patients
Anxiety visual analogic scales (VAS) | 30 minutes after using each interfaces
  evaluate the severity of anxiety the index has 10 numerical values, rated on a scale from 0-10, each value corresponding to an intensity pain and anxiety. It is an easy-to-use scale for patients
use of analgesic anti dyspnoetics drugs (morphine and derivatives) | 30 minutes after using each interfaces
  the type of molecule, dosage and route of administration will be identified
use of anxiolytic drugs | 30 minutes after using each interfaces
  the type of molecule, dosage and route of administration will be identified

CONTACTS AND LOCATIONS:
Overall Officials: Julie Delemazure, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.